CLINICAL TRIAL: NCT01682941
Title: Bioavailability of Isoflavones Delivered by Soy Almond Bread in Men With Recurring Prostate Cancer and Rising Prostate Specific Antigen
Brief Title: Soy Isoflavones in Treating Patients With Recurrent Prostate Cancer or Rising Prostate-Specific Antigen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yael Vodovotz, Associate Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OSU-08027; NCI-2010-02387 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA125909 (NIH)
Record Dates: First submitted 2012-09-06; First posted 2012-09-11 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Prostate Cancer; Stage IV Prostate Cancer
Keywords: soy, isoflavones, functional food, prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy Bread Intervention (Active Comparator): Arm I Soy Bread
  Interventions: Dietary Supplement: Arm I Soy Bread
- Soy -Almond Bread Intervention (Experimental): Arm II Soy-Almond Bread
  Interventions: Dietary Supplement: Arm II Soy-Almond Bread

INTERVENTIONS:
Dietary Supplement: Arm I Soy Bread — On day 0 or day 70 pharmacokinetic study of isoflavones over 24 hours will follow after consumption of 2 slices of soy bread. Afterwards 2 slices of soy bread/day will be consumed for 56 days and isoflavone metabolites will be assessed in urine at days 0, 28, 56, 70, 98, and 126.
  Other Names: soy isoflavones; soy phytoestrogens
  Arms: Soy Bread Intervention
Dietary Supplement: Arm II Soy-Almond Bread — On day 0 or day 70 pharmacokinetic study of isoflavones over 24 hours will follow after consumption of 2 slices of soy-almond bread. Afterwards 2 slices of soy-almond bread/day will be consumed for 56 days and isoflavone metabolites will be assessed in urine at days 0, 28, 56, 70, 98, and 126.
  Other Names: soy isoflavones; soy phytoestrogens
  Arms: Soy -Almond Bread Intervention

SUMMARY:
RATIONALE: Eating a diet high in soy foods may lower the risk of some types of cancer. Isoflavones are compounds found in soy food that may prevent cancer.

PURPOSE: This randomized phase II trial is studying how well soy isoflavones work in treating patients with recurrent prostate cancer or rising prostate-specific antigen

DETAILED DESCRIPTION:
OBJECTIVES:

I. To precisely quantify the absorption, serum concentrations over time, and excretion patterns of soy isoflavones and metabolites in men consuming the two bread products to define relationships between dietary intake, isoflavone metabolism and the biological outcomes.

II. To describe the safety as well as incidence and severity of toxicity in men consuming the control soy bread or beta-glucosidase-enriched soy bread.

III. To see if consumption of beta-glucosidase-enriched soy bread compared to control soy bread has a greater effect on blood hormonal patterns and biomarkers that favor anti-prostate cancer activity.

IV. To see if beta-glucosidase-enriched soy bread compared to control soy bread improves hormonal patterns (lower insulin like growth factor-I, increased insulin like growth factor binding protein 3, lower androgens), reduce prostate specific antigen velocity, and lower circulating vascular endothelial growth factor concentrations.

OUTLINE: Patients are randomized to 1 of 2 treatment arms (closed to accrual as of 02/14/2011).

ARM I: Patients consume 2 slices of soy bread daily for 8 weeks.

ARM II: Patients consume 2 slices of soy almond bread daily for 8 weeks.

After a 2 week washout period, patients crossover to the alternate treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed prostate cancer.
* Have completed primary therapy (radical prostatectomy, external beam radiation, brachytherapy) for prostate cancer. "Watchful waiting" patients will also be eligible.
* Have either two consecutive rises in prostate specific antigen (PSA) or a series of at least four PSA's over two years where the PSA doubling time is at least 3 months following a nadir response to localized therapy. The minimum PSA for this study is 0.2 ng/dL.
* Not be receiving ongoing chemotherapy, radiation therapy or biological therapy for internal malignancy including prostate cancer.
* At time of entry, the clinical team expects that no additional interventions for prostate cancer therapy (hormonal, chemotherapy, radiotherapy, etc.) will be necessary over the next 5 months.
* Not be currently using Finasteride, androgens, or other PSA modifying hormonal agents. Utilizing prescription medications for urinary outlet obstructive symptoms will not be permitted. The use of non-prescription substances to improve urinary tract symptoms will not be permitted (i.e. Saw Palmetto, other herbal, alternative products).
* Have kidney and liver enzymes within normal limits. Men with kidney and liver enzymes that are slightly elevated (< 1.5 times the upper normal limit), but have been stable for several months particularly those that are related to a known disorder (such as Gilberts syndrome, past history of alcohol, hepatitis, or a history of non-alcoholic steatohepatitis) will be permitted to participate after clinical evaluation by the study physician."
* Have no history of malabsorptive disorders or other metabolic disorders requiring special diet recommendations. Diabetics will be permitted to participate.
* Voluntarily agree to participate and a sign an informed consent document.
* Agree to consume a standardized vitamin and mineral supplement and avoid other nutrition, dietary, or alternative medications/supplements for the duration of the study.

Exclusion Criteria:

* Have an active malignancy other than prostate cancer that requires therapy.
* Have a history of pituitary hormone diseases that currently require supplemental hormonal administration (thyroid hormones, adrenocorticotropic hormone, growth hormone) or other endocrine disorders requiring hormone administration with the exception of diabetes, osteoporosis and men who have been stable (> 6 months of thyroid stimulating hormone within normal limits) on thyroid replacement therapy.
* Have a known allergy to tree nuts, soy or wheat protein.
* Have a recent history of iron deficient anemia (possible accentuation by soy).
* Antibiotic use in the last 6 months.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2015-06 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentrations (Cmax) of soy isoflavones and their metabolites | 0, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours post dose
  Quantification of absorption, serum concentrations over time, and excretion patterns of soy isoflavones and metabolites to define relationships between dietary intake, isoflavone metabolism and the biological outcomes

SECONDARY OUTCOMES:
Change in hormonal patterns after soy bread and soy-almond bread interventions | Day 0, 56, 70, and126
  Comparison of hormonal patterns (lower insulin like growth factor-I, increased insulin like growth factor binding protein-3, lower androgens), prostate specific antigen velocity, and circulating vascular endothelial growth factor concentrations
Changes in hormonal patterns that favor anti-prostate cancer activity | Days 0, 28, 56, 70, 98, and 126
  Comparison of isoflavone metabolites on blood hormonal patterns and biomarkers that favor anti-prostate cancer activity.
Severity of toxicity in participants after consumption of the control soy bread or beta-glucosidase-enriched soy almond bread | Day 0 and Day 126
  Safety (NIH criteria) and toxicity will be measured at day 0 (start of first intervention), day 56 (end of first intervention), day 70 (start of second intervention), and day 126 (end of second intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Vodovotz, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu